CLINICAL TRIAL: NCT05948501
Title: The Effects of Concussion on Gait and Posture in Individuals With Peripheral Vision Loss
Status: Withdrawn | Type: Observational
Why Stopped: Lack of resources to complete the study protocol as intended.
Sponsor: Gaylord Hospital, Inc (Other)
Collaborators: SOUTHERN CONNECTICUT STATE UNIVERSITY FOUNDATION INC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202303HRD
Record Dates: First submitted 2023-06-19; First posted 2023-07-17 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Concussion; Eye
Keywords: Concussion; Postural Control; Peripheral Vision Loss
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mTBI w/ Visual Impairment: Individuals 18 years or older, current patient of Gaylord Hospital Outpatient Services, within the last 6 months have been diagnosed with a mTBI/concussion with visual field loss of greater than or equal to 20% as determined by a perimetry screening
- mTBI w/o Visual Impairment: Individuals 18 years or older, current patient of Gaylord Hospital Outpatient Services, within the last 6 months have been diagnosed with a mTBI/concussion currently presenting with no symptoms consistent with peripheral vision loss.
- Healthy Control: Community dwelling adults aged 18 years or older with no diagnosis of mTBI/concussion within the last 6 months. Population will be matched to the concussion population within the age, gender, and height range of the concussion population.

SUMMARY:
Changes in gait and balance often occur in individuals who have suffered a concussion. In addition, a subset of concussed individuals also experience peripheral vision loss. To date, changes in gait and balance have not been examined in individuals who have suffered a concussion and also experience peripheral vision loss.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) results when an external force injures the brain and is a major cause of death and disability. In 2013 alone, an estimated 2.8 million people in the United States sustained a traumatic brain injury, most commonly from falls, being struck by or against an object, and motor vehicle accidents. The majority of traumatic brain injuries occur in patients aged 15-64 years during participation in sports. A frequent result of TBI is concussion caused by the rapid acceleration of the brain so that it impacts the inner walls of the skull which can cause both focal lesions such as cerebral laceration and hemorrhage and more diffuse damage resulting in edema and axonal injury. Retrospective studies show that 65 to 79% of patients with mild traumatic brain injury (mTBI) - a term often used interchangeably with concussion - report subjective visual complaints. The most common vision problems related to concussion include photophobia, visual processing problems, blurred vision, double vision and loss of vision (including decreased peripheral vision). For example, in 100 subjects 11-17 years of age with concussion, 69 percent had at least one visual problem, most commonly affecting accommodation, convergence, or saccadic and smooth pursuit movements. Also, in pediatric patients with concussion, 13 percent of 275 patients had persistent near point convergence abnormalities which were referred for vision therapy. The high frequency of visual involvement in concussion is not surprising, since more than half of the brain's pathways are dedicated to vision and eye movement control. The cognitive control of vision, in particular of eye movements, needs coordination of reflexive and voluntary activity, including frontoparietal circuits and subcortical nuclei; these pathways are vulnerable to injury in mTBI. While the topic of sports concussion has received a lot of media attention as a result of increased recognition of potential long-term deleterious effects of repeated concussive events, such as depression, altered cognition, and neurodegenerative diseases (e.g. chronic traumatic encephalopathy and Alzheimer's disease), the vision issues described above can also affect posture and balance. Postural control is essential to lead an independent life, perform activities of daily living, and ensure a correct gait.

Postural stability is maintained through the sensory integration of visual, vestibular, and proprioceptive inputs. The visual field is considered the most relevant visual function in falls. In humans, the visual field is divided into central vision (CV) and peripheral vision (PV). CV detects objects in the gaze direction, and PV detects the existence of surrounding objects, although imperfectly. There is some dispute in the literature as to the roles that central and peripheral visions play in maintaining balance. Three general hypotheses of visual field influences on postural control have been put forth in the literature: (1) the peripheral dominance theory is that peripheral vision is more important than central vision in postural control; (2) the retinal invariance hypothesis suggests that central vision is just as important as peripheral vision in the control of posture; and (3) the functional sensitivity hypothesis suggests that the periphery of the retina is most susceptible to lamellar optic flow and the central part is most sensitive to radial optic flow, and thus, both central and peripheral have important, but functionally different, roles in maintaining posture. Despite these three competing hypotheses of visual field influences on postural control, it is agreed upon that PV is closely related to postural control and sway and that those who have problems with PV have problems with postural control. Due to alterations in vestibular-visual feedback and sensorimotor control, individuals who have experienced a concussion frequently demonstrate gait abnormalities due to altered static and dynamic postural control. In addition to increased anterior-posterior (forward-backward) and medial-lateral (side-to-side) postural sway, concussed individuals have demonstrated decreases in gait velocity and step/stride length, wider step width, reduced cadence, and increased stance and double leg support time compared to normal, uninjured subjects. While the influence of PV loss on gait and posture has been studied in normal, healthy individuals, gait abnormalities in concussed individuals who have experienced PV loss has not been examined. Gait analysis has the benefit of detecting changes from a concussion that will be present after other criteria have been used to return individuals to participation. More specifically, there is preliminary evidence that gait deficits may exist beyond the typical 10-day recovery period and return to activity. Consensus about the most important gait parameters for concussion diagnosis and clinical management are lacking. Therefore, it is important to develop a better qualitative and quantitative understanding of changes in gait and posture in concussed individuals with PV loss. Analysis of gait may allow for the treatment of concussion patients to improve overall balance, movement efficiency, and overall quality of life.

ELIGIBILITY:
Inclusion Criteria; mTBI w/ Visual Impairment:

* Be 18 years of age or older.
* Be able to understand the study materials and provide informed consent.
* Be a current patient of Gaylord Hospital Outpatient Services.
* Within the last 6 months, have been diagnosed with a mild traumatic brain injury (mTBI)/concussion with visual field loss.
* Currently suffering symptoms consistent with peripheral vision loss.
* Have at least 20% vision loss as determined by a perimetry screening.
* Individuals with a history of one or more prior concussions that preceded the most recent mTBI may be included as long as the symptoms of the last concussion/mTBI had resolved prior to the most recent episode.
* Have completed 3 or fewer rehabilitation sessions prior to biomechanics testing.
* Ability to tolerate using the equipment required to complete the assessments for this study

Inclusion Criteria; mTBI w/o Visual Impairment

* Be 18 years of age or older.
* Be able to understand the study materials and provide informed consent.
* Be a current patient of Gaylord Hospital Outpatient Services
* Within the last 6 months, have been diagnosed with a mild traumatic brain injury (mTBI)/concussion without visual field loss
* Currently presenting with no symptoms consistent with peripheral vision loss.
* Have a perimetry no more than XX% vision loss as determined by perimetry screening.
* Individuals with a history of one or more prior concussions that preceded the most recent mTBI may be included as long as the symptoms of the last concussion/mTBI had resolved prior to the most recent episode.
* Have completed 3 or fewer rehabilitation sessions prior to biomechanics testing
* Ability to tolerate using the equipment required to complete the assessments for this study

Inclusion Criteria; Healthy Control

* Be a community dwelling adult 18 years of age or older.
* Be able to understand the study materials and provide informed consent.
* Have not experienced or been diagnosed with a concussion in the last 6 months
* Individuals with a history of one or more prior concussions, with or without vision loss, longer than 6 months prior to study recruitment may be considered as long as the symptoms of the last concussion/mTBI have resolved.
* Currently presenting with no symptoms consistent with peripheral vision loss.
* Have a perimetry no more than XX% vision loss as determined by perimetry screening.
* Ability to tolerate using the equipment required to complete the assessments for this study
* As this population will be matched to the concussion population, individuals must match fall within the age, gender, and height range of the concussion population

Exclusion Criteria:

* Moderate to severe TBI as diagnosed by imaging and physician diagnosis
* Participants who answer "YES" to any of the questions on the 2022 Physical Activities Readiness Questionnaire for Everyone (PAR-Q+)
* Current lower extremity injury
* Prior medical history or diagnosis that affects gait and/or balance
* Prior history of peripheral vision loss unrelated to current injury and diagnosis
* Peripheral neuropathy
* Pre-existing visual impairment not corrected by corrective lenses (glasses or contacts)
* Vestibular dysfunction (i.e. positional vertigo) that is unable to be cleared in 1 treatment session
* Cervicogenic range of motion limitations
* Any medical condition/medication that would interfere with subject safety or data collection in the opinion of the PI
* Member of a vulnerable or protected population, including people who are incarcerated, those under the age of 18, and those who are or might be pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include 3 populations of interest, a healthy control population, a population of individuals diagnosed with mTBI without visual impairment, and a population of individuals diagnosed with mTBI and subsequent visual impairment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Balance Test | This assessment will be collected upon enrollment in the study consisting of 1 day of testing. Outcome will be averaged across 3 trials.
  Static postural control test on a force plate (AMTI OR-6; Watertown, MA, USA).
Treadmill Walking Test | This assessment will be collected upon enrollment in the study consisting of 1 day of testing
  Participants will walk on an instrumented treadmill (Treadmetrix SDI; Park City, UT, USA) wearing their own comfortable shoes while their body segment motions will be recorded using an 8-camera markerless motion capture system (Theia Markerless, Inc., Kingston, ON, Canada) configured in an array around the perimeter of the treadmill. The treadmill walking test will utilize the Buffalo Concussion Treadmill Test (BCTT) protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Robert, Principal Investigator — Southern Connecticut University Foundation Inc; Henry Hrdlicka, PhD, Principal Investigator — Gaylord Specialty Healthcare
Locations (2):
- United States (2):
  - Southern Connecticut State University, New Haven, Connecticut
  - Gaylord Hospital, Wallingford, Connecticut

IPD SHARING:
Plan to Share IPD: No
Study was withdrawn prior to recruiting any participants and no participant data was collected as a result.